CLINICAL TRIAL: NCT07131813
Title: Evaluation of Efficacy and Safety of add-on Tofacitinib in Patients With Oral Lichen Planus: A Randomized Clinical Trial
Brief Title: Evaluation of Efficacy and Safety of add-on Tofacitinib in Patients With Oral Lichen Planus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/AIIMSBBSR/PGThesis/2025/46
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Oral Lichen Planus
Keywords: Tofacitinib; Oral Lichen Planus; Randomized Controlled Trial; Placebo; IL 6
MeSH Terms: conditions — Lichen Planus, Oral | interventions — tofacitinib; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The recruited patients were randomized into two treatment groups using block randomization (block size 6) with computer-generated random codes, maintaining an allocation ratio 1:1. Random allocation codes will be created by an investigator who does not participate in patient recruitment. The Sequentially Numbered, Opaque, Sealed Envelope (SNOSE) method will be employed to ensure allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Capsule Tofacitinib + Triamcinolone ointment (Experimental): Patients in the test group will get Tofacitinib 5mg twice daily as an add on to topical triamcinolone ointment
  Interventions: Drug: Tofacitinib 5 mg BID and Triamcinolone ointment
- Control: Placebo capsules + Triamcinolone ointment (Active Comparator): Patients in the control group will get similar looking capsules containing placebo in addition to triamcinolone ointment
  Interventions: Drug: Placebo and Triamcinolone ointment

INTERVENTIONS:
Drug: Tofacitinib 5 mg BID and Triamcinolone ointment — Patients in the test group will get tofacitinib 5mg capsules twice daily as an add on to triamcinolone ointment
  Arms: Test: Capsule Tofacitinib + Triamcinolone ointment
Drug: Placebo and Triamcinolone ointment — Patients in the control group will receive identical looking capsules as placebo with triamcinolone ointment
  Arms: Control: Placebo capsules + Triamcinolone ointment

SUMMARY:
Many of the patients with oral lichen planus (OLP) either fail to achieve complete remission or experience frequent relapses with conventional topical corticosteroid therapy, which is currently the mainstay of treatment. Long-term corticosteroid use is limited by local and systemic adverse effects, and many patients develop steroid resistance or intolerance. To overcome these limitations, combination therapy with agents having complementary mechanisms may improve therapeutic outcomes, reduce steroid requirements, and minimize associated adverse effects. Tofacitinib, a Janus kinase (JAK1/JAK3) inhibitor, modulates the JAK-STAT signaling pathway, thereby reducing inflammatory cytokine production involved in OLP pathogenesis. Preliminary case series and pilot trials have shown promising results with tofacitinib in OLP. However, to date, no randomized controlled trial has evaluated the efficacy and safety of add-on oral tofacitinib with standard topical steroid therapy in OLP. Hence, investigators considered tofacitinib to be a candidate drug for add-on therapy due to its anti-inflammatory and immunomodulatory properties. Adding tofacitinib to ongoing topical triamcinolone therapy may increase the response rate, reduce adverse drug reactions by lowering steroid dose requirements, or achieve a quicker therapeutic effect. Therefore, the present randomized controlled trial has been planned to evaluate the efficacy and safety of oral tofacitinib as an add-on therapy in patients with OLP.

DETAILED DESCRIPTION:
Lichen planus (LP) is a chronic, mucocutaneous inflammatory disorder that manifests as violaceous, polygonal, flat-topped papules and plaques, usually affecting the skin, oral mucosa, genital mucosa, and nails. Oral Lichen Planus (OLP) is the most persistent and symptomatic of its many forms, frequently impairing basic functions like eating, speaking, and swallowing. Oral Lichen Planus is an immune-mediated condition characterized by symmetrical, bilateral lesions most frequently seen on the tongue, gingiva, and buccal mucosa. Although the exact etiopathogenesis is unknown, antigen-specific T-cell-mediated cytotoxicity is thought to be a contributing factor. Early diagnosis, therapy, and follow-up are necessary because the disease has a relapsing-remitting course and, in a small percentage of patients, can potentially change into malignancies, particularly in its erosive and atrophic forms.

Oral Lichen Planus can be managed using a variety of treatment approaches, depending on its severity and clinical manifestation. Asymptomatic lesions can be controlled with observation and proper oral hygiene techniques without needing medication. Topical anesthetics and anti-inflammatory drugs can be used to treat mild cases of OLP. Because of their strong anti-inflammatory properties, topical corticosteroids continue to be the cornerstone of treatment for more severe atrophic or erosive forms. However, many patients have numerous relapses and are unable to attain complete remission with monotherapy. Adverse effects, such as oral candidiasis, mucosal thinning, and altered taste perception, are also linked to long-term usage of corticosteroids.

There is no definitive and proven treatment for OLP, despite the wide range of available options, including systemic immunosuppressants like cyclosporine and azathioprine and more recent techniques like laser therapy and photodynamic therapy. Furthermore, there aren't many well-designed, randomized controlled trials that direct standardized care. Therefore, the majority of therapy alternatives are empirical. Patients resistant to corticosteroids present a therapeutic dilemma, necessitating the exploration of newer, targeted options. Janus kinase (JAK) inhibitors, especially tofacitinib, have recently shown promise in treating immune-mediated dermatological disorders, including LP. Tofacitinib suppresses the generation of inflammatory cytokines associated with OLP pathogenesis by modulating the JAK-STAT signaling pathway through the selective inhibition of JAK1 and JAK3. According to preliminary case series and pilot trials, tofacitinib, when applied topically or systemically, can significantly improve erosive OLP, particularly in steroid-refractory cases.

However, to the best of investigator's knowledge, no randomized controlled trials have systematically evaluated the add-on effect of tofacitinib to standard topical steroid therapy in OLP patients. This represents a significant gap in current literature, particularly in defining the role of combination therapies that might offer enhanced efficacy, reduce cumulative steroid doses, and mitigate steroid-related adverse effects. Therefore, this study aims to evaluate the efficacy and safety of tofacitinib as an add-on to topical triamcinolone therapy in patients with oral lichen planus. This trial seeks to provide robust evidence that could potentially redefine treatment paradigms for OLP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 of either sex with the clinical diagnosis of oral lichen planus.
* Patients with a PGA score of ≥3 (moderate and severe oral LP).
* Patients who are willing to give informed written consent.

Exclusion Criteria:

* Treatment with a systemic corticosteroid within the last 4 weeks.
* Patients on immunosuppressive agents such as azathioprine, cyclosporine, and others within one month of recruitment.
* Patients with a clinical history and any lesion distribution suspicious of a lichenoid drug eruption, and patients with other skin diseases.
* Past or current history of any malignancy, including moderate to severe dysplasia of the oral mucosa on oral biopsy.
* Severe active infection, including active tuberculosis, hepatitis B, or C infection
* Patients with cytopenia (Hb <9g/dl, leukocyte count <4000/mm3, platelet count <100,000/mm3)
* The patient with a history of alcohol abuse.
* Decreased liver or renal function (creatinine > 2.0mg/dl, total bilirubin > 2.5 mg/dl).
* Severe acute infection, uncontrolled diabetes mellitus, congenital or acquired immunodeficiency, severe cardiac disease (NYHA grade IV), MI in the last four weeks, severe schizophrenia, or depression.
* Patient with a history of hypersensitivity to topical Triamcinolone or Tofacitinib.
* Pregnancy and lactation, women of childbearing age without effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in oral mucosal disease severity score from baseline | 4 weeks and12 weeks
  The change in oral mucosal disease severity score (maximum 106) will be evaluated using oral mucosal disease severity score questionnaire. Each item of the questionnaire yields a score of 0 to 106. A higher score depicts severe disease.

SECONDARY OUTCOMES:
Pain by Pain Visual Analogue Scale (VAS) score | 4 weeks and12 weeks
  Change in Pain Visual Analogue Scale (VAS) score after treatment with triamcinolone ointment and capsule tofacitinib vs. triamcinolone ointment and capsule placebo at baseline, 4 weeks, and 12 weeks. The VAS consists of a 10 cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Interpretation of the scores:0 = No pain, 2= Mild, 4 = Nagging, 6 = Miserable, 8 = intense, 10 = worst
Severity by Physician global assessment of disease (PGA) Score | 4 weeks and 12 weeks
  Compare the proportion of patients achieving a reduction of Physician Global Assessment of Disease (PGA) score of 0 or a 2-grade reduction (minimum initial PGA 3) after treatment with triamcinolone ointment and capsule tofacitinib vs. triamcinolone ointment and capsule placebo at baseline, 4 weeks, and 12 weeks by using a 6-point disease severity scoring system. (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, 5=very severe).
Quality of life by using oral health-related quality of life score (ORAL HEALTH IMPACT PROFILE - 14 ) | 4 weeks and 12 weeks
  Change in the oral health-related quality of life from baseline after 4 and 12 weeks. designed to assess patients' perception of the impact of oral disorders on their quality of life (QoL). The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse OHRQoL, and lower scores indicate better OHRQol
serum IL 6 level | 12 weeks
  Change in serum IL-6 after treatment with ointment triamcinolone and capsule tofacitinib vs. ointment triamcinolone and capsule placebo. The levels of salivary and serum IL-6 were significantly higher among patients with OLP than among healthy control participants
Incidence of treatment-emergent adverse events of both test and control group | 12 weeks
  treatment-emergent adverse events in both the groups The adverse events in the patients are to be assessed by non-directive questioning at the time of the follow-up visit. Patients can access the investigators directly in case of any adverse events and report them. All adverse events irrespective of their previous reported status are to be recorded with details about nature, intensity, duration, measures taken, outcome, and causal relationship to tofacitinib, triamcinolone and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Chair — Professor
Locations (1):
- AIIMS, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sandhu S, Klein BA, Al-Hadlaq M, Chirravur P, Bajonaid A, Xu Y, Intini R, Hussein M, Vacharotayangul P, Sroussi H, Treister N, Sonis S. Oral lichen planus: comparative efficacy and treatment costs-a systematic review. BMC Oral Health. 2022 May 6;22(1):161. doi: 10.1186/s12903-022-02168-4. PMID 35524296
- [Result] Kulkarni S, Durham H, Glover L, Ather O, Phillips V, Nemes S, Cousens L, Blomgran P, Ambery P. Metabolic adverse events associated with systemic corticosteroid therapy-a systematic review and meta-analysis. BMJ Open. 2022 Dec 22;12(12):e061476. doi: 10.1136/bmjopen-2022-061476. PMID 36549729
- [Result] Rotaru D, Chisnoiu R, Picos AM, Picos A, Chisnoiu A. Treatment trends in oral lichen planus and oral lichenoid lesions (Review). Exp Ther Med. 2020 Dec;20(6):198. doi: 10.3892/etm.2020.9328. Epub 2020 Oct 14. PMID 33123228
- [Result] Qing M, Yang D, Shang Q, Peng J, Deng J, Lu J, Li J, Dan H, Zhou Y, Xu H, Chen Q. CD8+ tissue-resident memory T cells induce oral lichen planus erosion via cytokine network. Elife. 2023 Aug 9;12:e83981. doi: 10.7554/eLife.83981. PMID 37555396
- [Result] Alrashdan MS, Cirillo N, McCullough M. Oral lichen planus: a literature review and update. Arch Dermatol Res. 2016 Oct;308(8):539-51. doi: 10.1007/s00403-016-1667-2. Epub 2016 Jun 27. PMID 27349424
- [Result] Katta R. Lichen planus. Am Fam Physician. 2000 Jun 1;61(11):3319-24, 3327-8. PMID 10865927